CLINICAL TRIAL: NCT05430568
Title: Comparison of Post-operation Cardiopulmonary Capacity of Patients Underwent Conventional and Robot-assisted Coronary Artery Bypass Graft and Valve Replacement Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CE22214A
Record Dates: First submitted 2022-05-29; First posted 2022-06-24 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Coronary Bypass Graft Stenosis; Valvular Heart Disease
Keywords: cardiorespiratory fitness; robotic assisted surgery; cardiopulmonary exercise testing
MeSH Terms: conditions — Heart Valve Diseases | interventions — Robotic Surgical Procedures; Sternotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- bypass graft, sternotomy: patients who have received coronary artery bypass graft surgery with conventional sternotomy procedure
- bypass graft, robot: patients who have received coronary artery bypass graft surgery with robot-assisted procedure
  Interventions: Procedure: robot-assisted surgery
- valvular heart disease, sternotomy: patients who have received valvular replacement surgery with conventional sternotomy procedure
- valvular heart disease, robot: patients who have received valvular replacement surgery with robot-assisted procedure
  Interventions: Procedure: robot-assisted surgery

INTERVENTIONS:
Procedure: robot-assisted surgery — 1. traditional sternotomy for coronary bypass graft or valvular replacement
  2. robot-assisted surgery for coronary bypass graft or valvular replacement
  Other Names: sternotomy
  Groups: bypass graft, robot; valvular heart disease, robot

SUMMARY:
Robotic surgery is one of the most popular minimally invasive procedures for patients with coronary artery disease or valvular diseases. Studies have shown that, as compared to conventional sternotomy, patients underwent robot-assisted bypass grafting or valvuloplasty had less post-operation pain, blood transfusion volume during operation, re-operation rate, post-operation stroke rate and length of hospitalization. However, most studies focused on the comparison of complications of different procedures, and the investigation of cardiopulmonary function recovery is still lacking. Thus our study is to compare the functional outcomes between patients that undergo different surgical procedures.

DETAILED DESCRIPTION:
The study is a prospective cohort study. The experimental group will include 40 patients, consisting 20 after robotic coronary artery bypass grafting and 20 after robotic valvuloplasty. The control group will include 20 patients for each conventional procedure.

Once decided the surgery type, the surgeon will consult the rehabilitation department and the director of this trial for inform consent. The recruitment and allocation will only be done after the patient has decided which type of surgery to receive. However, in case of change of surgery type, the patient will be excluded from the trial.

Cardiopulmonary exercise testing, 6-minute walking test and questionnaires about wound pain and cardiac functional status will be performed before surgery, two weeks after discharge and three months after discharge respectively. Primary outcomes include the change of maximal oxygen consumption (VO2), anaerobic threshold and the result of six minute walking test before and after surgery. Secondary outcomes include the change vital capacity (FVC), resting heart rate, oxygen pulse (O2 pulse), wound pain visual analog scale (VAS) and Duke Activity Status Index (DASI) before and after surgery.

The hypothesis of this study is that patients who undergo robot-assisted surgery will have better cardiopulmonary outcomes than those receive conventional surgery

ELIGIBILITY:
Inclusion Criteria:

* patient who undergo surgery for coronary artery bypass graft or valvular replacement.

Exclusion Criteria:

* pregnant
* patients who receive more than one type of surgery
* severe complications after surgery (ex. respiratory failure, stroke) and stayed in hospital for more than 2 weeks.
* cannot perform the cardiopulmonary exercise testing
* other contraindications for cardiopulmonary exercise testing

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: coronary artery and valvular heart disease patients
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Change of maximal oxygen consumption post-surgery | pre-operation to 2 weeks post-operation
  the change of maximal oxygen consumption from surgery before to 2 weeks after surgery
Change of maximal oxygen consumption in 3 months | pre-operation to 3 months post-operation
  the change of maximal oxygen consumption from before surgery to 3 months after surgery
Change of anaerobic threshold post surgery | pre-operation to 2 weeks post-operation
  the change of the onset of lactate accumulation in blood from before surgery to 2 weeks after surgery
Change of anaerobic threshold in 3 months | pre-operation to 3 months post-operation
  the change of the onset of lactate accumulation in blood from before surgery to 3 months after surgery
Change of six minute walking test result post-surgery | pre-operation to 2 weeks post-operation
  the change of six minute walking test result from before surgery to 2 weeks after surgery
Change of six minute walking test result in 3 months | pre-operation to 3 months post-operation
  the change of six minute walking test result from before surgery to 3 months after surgery

SECONDARY OUTCOMES:
Change of vital capacity post-surgery | pre-operation to 2 weeks post-operation
  the change of vital capacity during pulmonary function testing from before surgery to 2 weeks after surgery
Change of vital capacity in 3 months | pre-operation to 3 months post-operation
  the change of vital capacity during pulmonary function testing from before surgery to 3 months after surgery
Change of respiratory flow post-surgery | pre-operation to 2 weeks post-operation
  the change of the ratio of air volume on exhalation to vital capacity during the first second in the pulmonary function testing from before surgery to 2 weeks after surgery
Change of respiratory flow ratio in 3 months | pre-operation to 3 months post-operation
  the change of the ratio of air volume on exhalation to vital capacity during the first second in the pulmonary function testing from before surgery to 3 months after surgery
Change of resting heart rate post-surgery | pre-operation to 2 weeks post-operation
  the change of resting heart rate from before surgery to 2 weeks after surgery
Change of resting heart rate in 3 months | pre-operation to 3 months post-operation
  the change of resting heart rate from before surgery to 3 months after surgery
Change of oxygen pulse post-surgery | pre-operation to 2 weeks post-operation
  the change of the maximal value of VO2 divided by heart rate during exercise testing from before surgery to 2 weeks after surgery
Change of oxygen pulse in 3 months | pre-operation to 3 months post-operation
  the change of the maximal value of VO2 divided by heart rate during exercise testing from before surgery to 3 months after surgery
pain post-surgery | 2 weeks post-operation
  pain visual analog scale score (from 0 to 10, higher score means more painful) for surgery wound pain at 2 weeks after surgery
pain in 3 months | 3 months post-operation
  pain visual analog scale score (from 0 to 10, higher score means more painful) for surgery wound pain at 3 months after surgery
Change of activity status post-surgery | pre-operation to 2 weeks post-operation
  the change of the Duke Activity Status Index (DASI) score from before surgery to 2 weeks after surgery.
  The DASI is a score ranging from 0 to 58.2. A higher score indicates a better cardiorespiratory fitness.
Change of activity status in 3 months | pre-operation to 3 months post-operation
  the change of the Duke Activity Status Index (DASI) score from before surgery to 3 months after surgery The DASI is a score ranging from 0 to 58.2. A higher score indicates a better cardiorespiratory fitness.

CONTACTS AND LOCATIONS:
Overall Officials: Yuchun Lee, MD, Study Director — Taichung Veterans General Hospital
Locations (1):
- Department of Physical Medicine and Rehabilitation, Taichung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No